CLINICAL TRIAL: NCT04279938
Title: A Phase Ib Combination Study of Rituximab, TinostamustinEAnd CHeckpoint Inhibition With Pembrolizumab in Relapsed/Refractory DLBCL - REACH
Brief Title: A Phase Ib Combination Study of Rituximab, TinostamustinEAnd CHeckpoint Inhibition With Pembrolizumab in Relapsed/Refractory DLBCL
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety data on drug
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Mundipharma-EDO GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REACH - Trial Number pending
Record Dates: First submitted 2018-01-12; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Relapsed or Refractory Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, Large B-Cell, Diffuse | interventions — pembrolizumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safety Run in & Main Efficacy Part (Other): Part 1 (safety run-in) aims to evaluate the maximum tolerated dose (MTD) of tinostamustinein combination with pembrolizumab (200mg Q3W) and rituximab (375mg/m2 Q3W). The dose of tinostamustineestablished to be safe and tolerable in this combination will be used in part 2 of the trial (main efficacy part).
  The aim of part 2 is to detect signals of anti-tumour activity and to further assess the safety of this combination treatment in r/r DLBCL. The study has a strong focus on correlative research in order to identify mechanisms of response and resistance to pembrolizumab and the pembrolizumab/R-tinostamustinecombination.
  Interventions: Drug: Tinostamustinein; Drug: Pembrolizumab; Drug: Rituximab

INTERVENTIONS:
Drug: Tinostamustinein — Tinostamustine80-120mg IV Q3W (dose to be determined in part 1) for 6 cycles
Drug: Pembrolizumab — Pembrolizumab 200mg IV Q3W until disease progression or unacceptable toxicities (max. 2 years)
Drug: Rituximab — Rituximab 375 mg/m2 IV Q3W for 6 cycles

SUMMARY:
Safety run-in (part 1): Relapsed or refractory B-cell Non-Hodgkin lymphoma (NHL)

Main study (part 2): Relapsed or refractory diffuse large B-cell lymphoma

DETAILED DESCRIPTION:
The primary objective of the safety run-in phase (part 1) is to assess the safety and tolerability of pembrolizumab in combination with R-tinostamustineand to recommend a safe and tolerated dose of tinostamustinefor use in combination with 200mg pembrolizumab and 375mg/m2 rituximab Q3W in the main efficacy part of the study (part 2).

Part 2 (main study) The primary objective of part 2 is to assess efficacy of pembrolizumab in combination with R-tinostamustineas determined by the best overall response rate (ORR) in subjects with r/r DLBCL.

Hypothesis: The combination of pembrolizumab and R-tinostamustinewill act synergistically and show high anti-tumour efficacy in subjects with r/r DLBCL. R-EDO-S101 will increase pembrolizumab-mediated anti-tumour immunity by (A) tumour de-bulking with improved access of immune cells into the tumour and reduced burden of tumour sub-clones and (B) epigenetic priming of PD-1 inhibition through the histone deacetylase inhibitor (HDACi) component of tinostamustine.

Secondary Objectives & Hypotheses

1. Objective: Safety and tolerability of pembrolizumab in combination with R-tinostamustine.

   Hypothesis: Combination of pembrolizumab with R-tinostamustinewill be safe and well tolerated in r/r DLBCL patients.
2. Objective: Anti-tumour activity of pembrolizumab in combination with R-tinostamustineas determined by CR rate, duration of response (DOR), progression-free survival (PFS) and overall survival (OS).

Hypothesis: Combination of pembrolizumab with R-tinostamustinewill lead to deep and long remissions. Continuation of pembrolizumab treatment as maintenance after completion of induction therapy will demonstrate conversion of partial to complete response in some cases and prolonged stabilization of disease.

Exploratory Objectives

1. Objective: Minimal residual disease (MRD) detection in circulating cell-free tumour DNA (ctDNA) throughout treatment.

   Hypothesis: MRD assessment will enable better measurement of the depth of response in order to assess the effect of pembrolizumab after completion of R-tinostamustine/pembrolizumab induction.
2. Objective: Dynamics of circulating immune cell subsets in the peripheral blood (PB) throughout treatment.

   Hypotheses:
   * Detailed assessment of lymphocyte-, monocyte- and myeloid subsets and their protein expression from pre-treatment until disease progression will give insights into immunomodulation by pembrolizumab, and identify suitable pharmacodynamic markers and mechanisms of pembrolizumab resistance.
   * Assessment of PB T-cell function by synapse formation capacity and T-cell exhaustion will demonstrate restoration of T-cell defects by pembrolizumab.
3. Objective: Detailed analyses of tumour microenvironment (TME) changes during treatment and on progression.

   Hypotheses: Changes in the composition and function of tumour-associated immune- and stromal cells will elucidate mechanisms of action and resistance of pembrolizumab and the combination.
4. Objective: Evaluation of tumour-derived biomarkers of response and resistance. Hypotheses: Association of the molecular background of DLBCL (somatic mutations, mRNA and protein expression, DNA methylation) with treatment response will help to identify predictive biomarkers for future validation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven CD20+ DLBCL (including transformed lymphoma)
* Previous treatment with at least 1 line of standard therapy
* Age 18 or over
* ECOG performance status 0/1 Measurable disease on cross-sectional imaging that is at least 1.5 cm in the longest diameter and measureable in two perpendicular dimensions
* Adequate organ function
* Resolution of prior systemic therapy related non-haematological AEs to grade (G) ≤ 1. Participants with ≤ G 2 neuropathy may be eligible.
* Consent to provide fresh tumour tissue during screening and treatment

Exclusion Criteria:

* CNS or leptomeningeal involvement
* Autologous stem cell transplant (ASCT) within 12 weeks or other anticancer treatment within 3 weeks of commencing therapy
* Prior allogeneic transplant
* Known HIV, or active Hepatitis B/C infection
* Active systemic autoimmune disease
* No previous therapy with agents targeting immune checkpoint proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2.3 years
  Part 1 (safety run-in): To assess the safety and tolerability of pembrolizumab in combination with R-tinostamustineand to recommend a safe and tolerated dose of tinostamustinefor use in part 2 in combination with 200mg pembrolizumab and 375mg/m2 rituximab .
  Part 2 (main study): To assess efficacy of pembrolizumab in combination with R-tinostamustineas determined by best overall response in subjects with relapsed/refractory (r/r) DLBCL.

SECONDARY OUTCOMES:
Secondary Objectives | 2.3 years
  Anti-tumour activity of pembrolizumab in combination with R-tinostamustineas determined by complete response rate (CR), duration of response (DOR), progression-free survival (PFS) and overall survival (OS)
  * To assess the safety profile of pembrolizumab in combination with R-tinostamustinein subjects with r/r DLBCL
  * Exploratory biomarkers of response and resistance to pembrolizumab in combination with R-tinostamustine

CONTACTS AND LOCATIONS:
Overall Officials: Professor David Cunningham, Study Chair — The Royal Marsden Hospital NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No